CLINICAL TRIAL: NCT05504811
Title: FitMi AD: a Safe and Motivating Computer-guided Exercise System for Individuals With MCI or Mild Dementia Due to Alzheimer's Disease
Brief Title: FitMi AD Home Therapy for Individuals With MCI or Mild Dementia Due to Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flint Rehabilitation Devices, LLC (Industry)
Collaborators: Rancho Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2R44AG063651-02 (NIH)
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Dysfunction; Dementia, Mild
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental: FitMi AD Exercise Program (Experimental): Participants will perform exercises by interacting with FitMi pucks, as described and monitored on a tablet computer. Participants will be asked to exercise at least 30 minutes per day for 3 months.
  Interventions: Device: FitMi AD
- Active Comparator: Conventional booklet of exercise program (Active Comparator): Participants will perform exercises described in a booklet similar to what is typically provided to individuals. Participants will be asked to exercise at least 30 minutes per day for 3 months.
  Interventions: Other: Conventional exercise program

INTERVENTIONS:
Device: FitMi AD — Exercise using the motion sensing devices and a tablet computer
  Arms: Experimental: FitMi AD Exercise Program
Other: Conventional exercise program — Exercise following printed sheets or booklet
  Arms: Active Comparator: Conventional booklet of exercise program

SUMMARY:
This study will investigate the efficacy of a newly developed exercise device (FitMi AD) for individuals with mild cognitive impairment (MCI) or mild dementia due to Alzheimer's disease. FitMi AD uses embedded sensors that can track and record the patient's direction and degree of movement while performing exercises described on a computer.

ELIGIBILITY:
Inclusion Criteria:

* have MCI or mild dementia due to AD (i.e. Clinical Dementia Rating (CDR) score 1 for mild dementia or 0.5 for MCI)
* ability to clearly see the screen and hear the audio instructions from the tablet
* have a family member or friend who can answer questions about the participant's daily living skills
* willing to participate in a research study.

Exclusion Criteria:

* age < 50 years old
* use of a wheelchair as a primary mobility device (use of a cane or walker is permitted)
* presence of other neurologic conditions such as movement disorders or history of stroke
* other severe concurrent medical conditions that may prevent the participants from completing the 3-month study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Change in Functional Reach Test | Baseline, Immediately Post-Treatment (an average of 3 months)
  How far can someone reach while standing in a fixed position
Change in Timed Up and Go test | Baseline, Immediately Post-Treatment (an average of 3 months)
  Time it takes to stand up from a chair and walk a short distance
Change in 30 second chair stand test | Baseline, Immediately Post-Treatment (an average of 3 months)
  How many times someone stand up from a chair in 30 seconds

SECONDARY OUTCOMES:
Visual Analog Pain Scale | Baseline, Immediately Post-Treatment (an average of 3 months)
  Indicates perceived pain intensity. The scale consists of a line, often 10 cm long, with verbal anchors at either end (i.e. "no pain" on the far left and "the most intense pain imaginable" on the far right). The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity.
Global Physical Activity Questionnaire | Baseline, Immediately Post-Treatment (an average of 3 months)
  Assesses physical activity habits
Geriatric Depression Scale | Baseline, Immediately Post-Treatment (an average of 3 months)
  Evaluates depression in elderly individuals. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Pittsburgh Sleep Quality Index | Baseline, Immediately Post-Treatment (an average of 3 months)
  Measures the quality and patterns of sleep in adults. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Duration of exercise performed | Immediately Post-Treatment (an average of 3 months)
  Duration of exercise performed over intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Freddi Segal-Gidan, PA, PhD, Principal Investigator — Rancho Research Institute, Inc.
Locations (1):
- Rancho Research Institute, Inc, Downey, California, United States